CLINICAL TRIAL: NCT00004913
Title: A Phase I Study of Docetaxel Plus 5-FU, Cisplatin and Leucovorin in Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 98X2; NU-98X2; NCI-G00-1707
Record Dates: First submitted 2000-03-07; First posted 2004-03-16 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Docetaxel; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of docetaxel administered in combination with cisplatin, fluorouracil, and leucovorin calcium in patients with advanced solid tumors. II. Determine the toxicities associated with this combination regimen in this patient population. III. Evaluate the clinical response to this combination regimen in these patients.

OUTLINE: This is a dose escalation study of docetaxel and fluorouracil (5-FU). Patients receive docetaxel IV over 1 hour on day 1, cisplatin IV over 1 hour on day 2, and leucovorin calcium IV immediately followed by 5-FU IV on days 1-5. Treatment repeats every 3 weeks in the absence of disease progression. Cohorts of 3-5 patients receive escalating doses of docetaxel and 5-FU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which more than 1 of 3 or 1 of 5 patients experience dose limiting toxicity. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of advanced solid tumor No lymphomas Measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AND SGOT no greater than 2.5 times ULN AND Alkaline phosphatase no greater than ULN OR SGOT no greater than ULN AND Alkaline phosphatase no greater than 5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: No pre-existing peripheral neuropathy greater than grade 2 Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: No more than 2 prior treatments for metastatic disease Biologic therapy: Not specified Chemotherapy: No prior high dose (pre transplant) chemotherapy Prior paclitaxel allowed Endocrine therapy: Not specified Radiotherapy: No prior pelvic radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al B. Benson, MD, FACP, Study Chair — Robert H. Lurie Cancer Center
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania